CLINICAL TRIAL: NCT01064297
Title: Lamotrigine Pregnancy Registry (LAM05)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112913; 105905 (Other: GSK); EPI40048 (Other: GSK)
Record Dates: First submitted 2010-01-28; First posted 2010-02-08 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Epilepsy; Bipolar Disorder
Keywords: Pregnancy registry; Major congenital malformations; Pregnancy outcomes; Pregnancy; First trimester; Lamotrigine
MeSH Terms: conditions — Epilepsy; Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women exposed to lamotrigine during pregnancy
  Interventions: Drug: Lamotrigine monotherapy; Drug: Lamotrigine polytherapy including valproate; Drug: Lamotrigine polytherapy without valproate

INTERVENTIONS:
Drug: Lamotrigine monotherapy — Lamotrigine monotherapy
Drug: Lamotrigine polytherapy including valproate — Lamotrigine polytherapy including valproate
Drug: Lamotrigine polytherapy without valproate — Lamotrigine polytherapy without valproate

SUMMARY:
Antiepileptic drugs (AEDs) are not indicated for use in pregnancy. However, women with epilepsy, and other approved indications including bipolar disorder, may require or be unintentionally exposed to AEDs during pregnancy. Prior to an AED being marketed there are few data available on drug safety in pregnancy: data from animal models may not translate directly to humans and pregnant women are routinely excluded from clinical trials. The International Lamotrigine Pregnancy Registry was established by GlaxoSmithKline (GSK) in 1992 to monitor the safety of lamotrigine during pregnancy.

DETAILED DESCRIPTION:
The International Lamotrigine Pregnancy Registry aims to assess whether there is a substantial increase in the risk of major congenital malformations (MCMs) following in utero exposure to lamotrigine. Exposure during the first trimester is of primary interest as this represents the period of organogenesis. The Registry is a primarily prospective enrolment and follow-up study. Patients exposed to lamotrigine during pregnancy are enrolled, on a voluntary basis, by their healthcare provider. Enrolment is encouraged early in pregnancy and if possible prior to any prenatal testing. The healthcare provider provides initial information concerning patient demographics; details of the pregnancy including the estimated delivery date and results of any prenatal testing; and the timing, duration and dosage of lamotrigine exposure in pregnancy. The registry accepts exposure reports from anywhere in the world. Within the United States (US) the healthcare provider can contact the registry using a toll free number. Outside of the US enrolments are made through the GlaxoSmithKline local operating company.

Close to the estimated date of delivery the healthcare provider is contacted by the Registry to provide follow up information concerning the pregnancy outcome (live or still birth, spontaneous or induced abortion), the presence or absence of a MCM, and the history of exposure to lamotrigine as well other antiepileptics and antipsychotics during pregnancy. Up to six attempts are made to contact the healthcare provider to obtain pregnancy outcome information. After six attempts, the record is closed as lost to follow up. Pregnancy outcomes are classified as outcomes with MCMs, outcomes without MCMs and spontaneous abortions. The outcomes with and without MCMs are further classified as live births, stillbirths/fetal deaths and induced abortions. Spontaneous abortions are reported separately due to potential for inconsistent identification of malformations in that situation.

It is beyond the scope of the Registry to consistently access pediatric evaluations and medical records. For this reason the main outcome is restricted to major congenital malformations that are external and recognizable in the delivery room or shortly after birth. To provide consistency, reported congenital malformations are classified as major or minor according to criteria used by the Centers for Disease Control and Prevention (CDC)'s Metropolitan Atlanta Congenital Defects Program (MACDP). All malformation reports are reviewed and classified by a paediatrician from the CDC and further information is requested as necessary.

Analyses are restricted to prospectively enrolled pregnancies (enrolment prior to knowledge of the birth outcome). Retrospectively enrolled pregnancies are reviewed for patterns of defect types, but are not included in formal analyses as retrospective reporting can be biased towards more unusual and severe outcomes and are less likely to be representative of the general population experience. The proportion of infants with MCMs among prospectively reported exposures is calculated as: the total number of outcomes with major birth defects (number of outcomes with major birth defects + the number of live births without defects).

Chromosomal malformations are reported descriptively, but are not included in the numerator as it is very unlikely that they are associated with drug exposure during pregnancy. All spontaneous pregnancy losses, as well as induced abortions and fetal deaths without reported defects, are excluded from the denominator due to the potential for inconsistent identification of malformations in those situations. The 95% confidence intervals (CIs) for risk estimates are calculated using exact methods based on the binomial distribution.

Analyses are stratified according to trimester of exposure (with the second trimester starting at week 14 and the third trimester at week 28 of gestation) and by exposure group (lamotrigine monotherapy, lamotrigine polytherapy including valproate and lamotrigine polytherapy without valproate).

The registry does not have an internal comparator group, but descriptive comparisons are made with MCM rates from general population studies in the literature and from other ongoing AED pregnancy registries. Prospective reports are also reviewed to detect any unusual patterns of malformation types that may warrant further investigation. The data from the International Lamotrigine Pregnancy Registry are reviewed, and conclusions developed, by an independent scientific advisory committee. A semi-annual interim report summarizing aggregate data is provided to disseminate information on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Women exposed in utero to lamotrigine (as monotherapy or in a polytherapy combination) during pregnancy. Exposure can occur at any time during pregnancy, though exposure in the first trimester is of primary interest.
* Pregnancies exposed to lamotrigine and reported before the outcome of the pregnancy is known (prospective reporting). Ideally exposed pregnancies are registered prior to prenatal testing, but only those pregnancies enrolled after prenatal testing has diagnosed a birth defect are excluded.
* Retrospectively reported exposures (i.e. exposures registered once the pregnancy outcome is known) are included in the registry, but are considered descriptively and are not included in risk analyses.

Exclusion Criteria:

* Retrospectively reported exposures (i.e. exposures registered once the pregnancy outcome is known) are included in the registry, but are reviewed separately and descriptively. These are not included in risk analyses.
* Patient reported exposures and outcomes that are not verified by a healthcare provider.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to lamotrigine during pregnancy anywhere in the world.
Sampling Method: Non-Probability Sample
Enrollment: 3416 (Actual)
Dates: Start 2001-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Cunnington MC, Weil JG, Messenheimer JA, Ferber S, Yerby M, Tennis P. Final results from 18 years of the International Lamotrigine Pregnancy Registry. Neurology. 2011 May 24;76(21):1817-23. doi: 10.1212/WNL.0b013e31821ccd18. PMID 21606453
- [Background] Cunnington M, Ferber S, Quartey G; International Lamotrigine Pregnancy Registry Scientific Advisory Committee. Effect of dose on the frequency of major birth defects following fetal exposure to lamotrigine monotherapy in an international observational study. Epilepsia. 2007 Jun;48(6):1207-10. doi: 10.1111/j.1528-1167.2007.01021.x. Epub 2007 Mar 22. PMID 17381445
- [Background] Cunnington M, Tennis P; International Lamotrigine Pregnancy Registry Scientific Advisory Committee. Lamotrigine and the risk of malformations in pregnancy. Neurology. 2005 Mar 22;64(6):955-60. doi: 10.1212/01.WNL.0000154515.94346.89. PMID 15781807
- [Background] Cunnington MC. The International Lamotrigine pregnancy registry update for the epilepsy foundation. Epilepsia. 2004 Nov;45(11):1468. doi: 10.1111/j.0013-9580.2004.451105.x. No abstract available. PMID 15509254
- [Background] Lamotrigine Pregnancy Registry. Interim Report 1 September 1992 through 31 March 2010. Issued July 2010. Available at: http://pregnancyregistry.gsk.com/index.html
- [Background] Tennis P, Eldridge RR; International Lamotrigine Pregnancy Registry Scientific Advisory Committee. Preliminary results on pregnancy outcomes in women using lamotrigine. Epilepsia. 2002 Oct;43(10):1161-7. doi: 10.1046/j.1528-1157.2002.45901.x. PMID 12366730

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine Monotherapy Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine monotherapy at doses between 0-1200 mg/day
- Lamotrigine Polytherapy With Valproate Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine polytherapy with valproate, all dose ranges
- Lamotrigine Polytherapy Without Valproate Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine polytherapy without valproate, all dose ranges
Period: Overall Study
Arm/Group | Lamotrigine Monotherapy Pregnancy Exposures | Lamotrigine Polytherapy With Valproate Pregnancy Exposures | Lamotrigine Polytherapy Without Valproate Pregnancy Exposures
Started | 2567 | 219 | 630
Completed | 1776 | 171 | 497
Not Completed | 791 | 48 | 133
Not completed — Lost to Follow-up | 791 | 48 | 133

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine Monotherapy Pregnancy Exposures | Lamotrigine Polytherapy With Valproate Pregnancy Exposures | Lamotrigine Polytherapy Without Valproate Pregnancy Exposures | Total
Number analyzed (Participants) | 2567 | 219 | 630 | 3416
Age Continuous [Mean (Standard Deviation); unit: years] — Prospectively enrolled pregnancies with pregnancy outcome known or lost to follow-up.
  years | 27.9 (5.84) | 25.8 (5.49) | 28.1 (6.08) | 27.8 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants] — Prospectively enrolled pregnancies with pregnancy outcome known or lost to follow-up.
  Participants
    Female | 2567 | 219 | 630 | 3416
    Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Birth Outcomes by Earliest Pregnancy Trimester of Exposure to Lamotrigine Monotherapy
Description: The number of live births, fetal deaths, induced abortions, and spontaneous pregnancy losses were recorded according to the time at which women were first exposed to lamotrigine monotherapy. Due to inconsistent identification of major congenital malformations (MCMs) among spontaneous losses, no comment is made concerning the presence or absence of MCMs.
Time Frame: Although reports and diagnoses of major congenital malformations are accepted up to six years after the birth, the majority of malformations are reported after assessments made in the delivery room or shortly after birth
Population: Prospectively enrolled pregnancies exposed to lamotrigine monotherapy.
Measure: Number; unit: infants
Groups:
- First Exposure During First Trimester: The first trimester begins at conception
- First Exposure During Second Trimester: The second trimester begins at 14 weeks gestation
- First Exposure During Third Trimester: The third trimester begins at 28 weeks gestation
- Unspecified Trimester of Exposure: The earliest trimester of exposure was not specified
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure
Number analyzed (Participants) | 1699 | 95 | 18 | 5
infants
  Live Birth (Birth Defects Reported) | 31 | 4 | 1 | 0
  Fetal Death (Birth Defects Reported) | 1 | 0 | 0 | 0
  Induced Abortion (Birth Defects Reported) | 3 | 0 | 0 | 0
  Live Birth (No Birth Defects Reported) | 1523 | 91 | 17 | 5
  Fetal Death (No Birth Defects Reported) | 10 | 0 | 0 | 0
  Induced Abortion (No Birth Defects Reported) | 33 | 0 | 0 | 0
  Spontaneous Pregnancy Loss | 98 | 0 | 0 | 0

2. Primary Outcome: Birth Outcomes by Earliest Pregnancy Trimester of Exposure to Lamotrigine Polytherapy With Valproate
Description: The number of live births, fetal deaths, induced abortions, and spontaneous pregnancy losses were recorded according to the time at which women were first exposed to lamotrigine polytherapy with valproate. Due to inconsistent identification of major congenital malformations (MCMs) among spontaneous losses, no comment is made concerning the presence or absence of MCMs.
Time Frame: Although reports and diagnoses of MCMs are accepted up to six years after the birth, the majority of malformations are reported following assessments made in the delivery room or shortly after birth
Population: Prospectively enrolled pregnancies exposed to lamotrigine polytherapy with valproate.
Measure: Number; unit: infants
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure
Number analyzed (Participants) | 161 | 8 | 3 | 1
infants
  Live Birth (Birth Defects Reported) | 14 | 1 | 0 | 0
  Fetal Death (Birth Defects Reported) | 0 | 0 | 0 | 0
  Induced Abortion (Birth Defects Reported) | 2 | 0 | 0 | 0
  Live Birth (No Birth Defects Reported) | 134 | 6 | 3 | 1
  Fetal Death (No Birth Defects Reported) | 1 | 1 | 0 | 0
  Induced Abortion (No Birth Defects Reported) | 4 | 0 | 0 | 0
  Spontaneous Pregnancy Loss | 6 | 0 | 0 | 0

3. Primary Outcome: Birth Outcomes by Earliest Pregnancy Trimester of Exposure to Lamotrigine Polytherapy Without Valproate
Description: The number of live births, fetal deaths with pregnancy loss occurring >=20 weeks gestation, induced abortions, and spontaneous pregnancy losses were recorded according to the time at which women were first exposed to lamotrigine polytherapy without valproate. Due to inconsistent identification of major congenital malformations (MCMs) among spontaneous losses, no comment is made concerning the presence or absence of MCMs. Although birth defects may not have been reported, they cannot be ruled out.
Time Frame: as for outcome 2
Population: Prospectively enrolled pregnancies exposed to the lamotrigine polytherapy without valproate
Measure: Number; unit: infants
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure
Number analyzed (Participants) | 474 | 25 | 3 | 0
infants
  Live Birth (Birth Defects Reported) | 11 | 0 | 1 |
  Fetal Death (Birth Defects Reported) | 0 | 0 | 0 |
  Induced Abortion (Birth Defects Reported) | 1 | 0 | 0 |
  Live Birth (No Birth Defects Reported) | 418 | 25 | 2 |
  Fetal Death (No Birth Defects Reported) | 3 | 0 | 0 |
  Induced Abortion (No Birth Defects Reported) | 19 | 0 | 0 |
  Spontaneous Pregnancy Loss | 22 | 0 | 0 |

4. Primary Outcome: Number of Infants With Major Congenital Malformations by Earliest Trimester of Exposure to Lamotrigine Monotherapy
Description: Among lamotrigine monotherapy exposures: live births, fetal deaths, induced abortions with birth defects, and live births without defects. Due to the likelihood of inconsistent identification of birth defects among spontaneous losses, fetal deaths, and induced abortions without reported birth defects, these offspring were not included in analyses.
Time Frame: Although reports and diagnoses of MCMs are accepted up to six years after the birth, the majority of malformations are reported after assessments made in the delivery room or shortly after birth
Population: Among lamotrigine monotherapy exposures: live births, fetal deaths, induced abortions with birth defects, and live births without defects. Due to the likelihood of inconsistent identification of birth defects among spontaneous losses, fetal deaths, and induced abortions without reported birth defects, these offspring were not included in analyses.
Measure: Number; unit: infants
Groups:
- All Trimesters: Exposure during any trimester of pregnancy
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure | All Trimesters
Number analyzed (Participants) | 1558 | 95 | 18 | 5 | 1676
infants | 35 | 4 | 1 | 0 | 40
Statistical Analysis 1: Comparison: First Exposure During First Trimester; Test type: Superiority or Other; Wilson Score with Continuity Correction = 2.2, 95% CI [1.6 to 3.1] — The percentage of infants with MBDs was calculated as: the number of outcomes with MBDs divided by (the number of outcomes with MBDs + the number of live births without defects)
Statistical Analysis 2: Comparison: First Exposure During Second Trimester; Test type: Superiority or Other; Wilson Score with Continuity Correction = 4.2, 95% CI [1.4 to 11.0] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: All Trimesters; Test type: Superiority or Other; Wilson Score with Continuity Correction = 2.4, 95% CI [1.7 to 3.3] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Number of Infants With Major Congenital Malformations (MCMs) by Earliest Trimester of Exposure to Lamotrigine Polytherapy With Valproate
Description: The number of infants with major congenital malformations were counted and are presented by earliest trimester of exposure to lamotrigine polytherapy with valproate.
Time Frame: as for outcome 2
Population: Among lamotrigine polytherapy with valproate exposures: live births, fetal deaths, induced abortions with defects, and live births without defects. Due to the likelihood of inconsistent identification of defects among spontaneous losses, fetal deaths, and induced abortions without reported defects, these offspring were not included in analyses.
Measure: Number; unit: infants
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure | All Trimesters
Number analyzed (Participants) | 150 | 7 | 3 | 1 | 161
infants | 14 | 1 | 0 | 0 | 1
Statistical Analysis 1: Comparison: First Exposure During First Trimester; Test type: Superiority or Other; Wilson Score with Continuity Correction = 10.7, 95% CI [6.4 to 17.0]
Statistical Analysis 2: Comparison: All Trimesters; Test type: Superiority or Other; Wilson Score with Continuity Correction = 9.3, 95% CI [5.5 to 15.2] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Number of Infants With Major Congenital Malformations (MCMs) by Earliest Trimester of Exposure to Lamotrigine Polytherapy Without Valproate
Description: The number of infants with major congenital malformations were counted and are presented by earliest trimester of exposure to lamotrigine polytherapy without valproate.
Time Frame: as for outcome 2
Population: Among lamotrigine polytherapy without valproate exposures: live births, fetal deaths, induced abortions with defects, and live births without defects. Due to the likelihood of inconsistent identification of defects among spontaneous losses, fetal deaths, and induced abortions without reported defects, these offspring were not included in analyses.
Measure: Number; unit: infants
Arm/Group | First Exposure During First Trimester | First Exposure During Second Trimester | First Exposure During Third Trimester | Unspecified Trimester of Exposure | All Trimesters
Number analyzed (Participants) | 430 | 25 | 3 | 0 | 458
infants | 12 | 0 | 1 |  | 13
Statistical Analysis 1: Comparison: First Exposure During First Trimester; Test type: Superiority or Other; Wilson Score with Continuity Correction = 2.8, 95% CI [1.5 to 5.0]
Statistical Analysis 2: Comparison: All Trimesters; Test type: Superiority or Other; Wilson Score with Continuity Correction = 2.8, 95% CI [1.6 to 4.9] — [estimate comment as in outcome 4, analysis 1]

7. Primary Outcome: Number of Infants With the Indicated Major Congenital Malformations Following the First Trimester of Exposure to Lamotrigine Monotherapy According to Dose Received
Description: The number of infants with the reported MCM following first trimester lamotrigine monotherapy exposure were counted. Registry personnel contacted the enrolling physician to obtain information on the pregnancy outcome, lamotrigine dosing and duration of exposure, and use of concomitant antiepileptic drugs during pregnancy.
Time Frame: as for outcome 4
Population: Among lamotrigine monotherapy exposures in the first trimester: live births, fetal deaths, induced abortions with defects, and live births without defects. Due to the likely inconsistent identification of defects among spontaneous losses, fetal deaths, and induced abortions without reported defects, these offspring were not included in analyses.
Measure: Number; unit: infants
Groups:
- Doses Lower Than Prescribed: >0 to 200 mg/day maximal dose in first trimester
- Prescribed Doses: 201-400 mg/day maximal dose in first trimester
- Dose Higher Than Prescribed: >400 mg/day maximal dose in first trimester
Arm/Group | Doses Lower Than Prescribed | Prescribed Doses | Dose Higher Than Prescribed | Unknown Maximal Dose in Exposed Trimester
Number analyzed (Participants) | 15 | 12 | 6 | 2
infants
  Anencephaly | 2 | 0 | 1 | 0
  Orofacial clefts | 2 | 0 | 0 | 0
  Hypoplastic left heart/left ventricle hypoplasia | 1 | 0 | 1 | 0
  Transposition of great vessels | 2 | 0 | 0 | 0
  Ventricular septal defects | 0 | 3 | 0 | 0
  Minor heart defect, unspecified | 0 | 1 | 0 | 0
  Pulmonary stenosis | 0 | 1 | 0 | 0
  Hydronephrosis | 1 | 1 | 0 | 0
  Renal defect (absent, polysystic, fluid on kidney) | 1 | 0 | 2 | 0
  Cortical dysplasis | 0 | 1 | 0 | 0
  Hypospadias | 1 | 1 | 0 | 0
  Pyloric stenosis | 0 | 1 | 0 | 1
  Diaphragmatic hernia | 1 | 0 | 1 | 0
  Congenital atresia of anus | 1 | 0 | 0 | 0
  Hip dislocation | 1 | 0 | 0 | 0
  Club feet | 0 | 1 | 1 | 1
  Polydactyly | 1 | 1 | 0 | 0
  Epidermolysis bullosa | 1 | 0 | 0 | 0
  Light spot across entire abdomen | 0 | 1 | 0 | 0

8. Primary Outcome: Number of Infants With the Indicated Major Congenital Malformations Following First Trimester of Exposure to Lamotrigine Polytherapy With Valproate According to Dose of Lamotrigine Received
Description: The number of infants with the reported MCM following first trimester exposure to lamotrigine polytherapy with valproate were counted.
Time Frame: as for outcome 4
Population: Among lamotrigine polytherapy with valproate exposures in the first trimester: live births, fetal deaths, induced abortions with defects, and live births without defects. Due to the likely inconsistent identification of defects among spontaneous losses, fetal deaths, and induced abortions without reported defects, those offspring were excluded.
Measure: Number; unit: infants
Groups:
- Doses Higher Than Prescribed: >400 mg/day maximal dose in first trimester
Arm/Group | Doses Lower Than Prescribed | Prescribed Doses | Doses Higher Than Prescribed | Unknown Maximal Dose in Exposed Trimester
Number analyzed (Participants) | 13 | 3 | 0 | 0
infants
  Hydrocephalus/spina bifida | 1 | 0 |  |
  Meningomyelocele | 1 | 0 |  |
  Microcephaly | 1 | 0 |  |
  Orofacial clefts | 2 | 1 |  |
  Cardiac septal defects | 0 | 2 |  |
  Transposition of great vessels | 1 | 0 |  |
  Ventricular hypoplasia | 1 | 0 |  |
  Pulmonary stenosis | 1 | 0 |  |
  Pyloric stenosis | 1 | 0 |  |
  Gastroschisis | 1 | 0 |  |
  Club foot | 2 | 0 |  |
  Polydactyly | 1 | 0 |  |

9. Primary Outcome: Number of Infants With the Indicated Major Congenital Malformations Following First Trimester of Exposure to Lamotrigine Polytherapy Without Valproate According to Dose of Lamotrigine Received
Description: The number of infants with the reported MCM following first trimester exposure to lamotrigine polytherapy without valproate were counted.
Time Frame: as for outcome 4
Population: Among lamotrigine polytherapy without valproate exposures in the first trimester: live births, fetal deaths, induced abortions with defects, and live births without defects. Due to the likely inconsistent identification of defects among spontaneous losses, fetal deaths, and induced abortions without reported defects, those offspring were excluded.
Measure: Number; unit: infants
Arm/Group | Doses Lower Than Prescribed | Prescribed Doses | Doses Higher Than Prescribed | Unknown Maximal Dose in Exposed Trimester
Number analyzed (Participants) | 2 | 4 | 6 | 0
infants
  Neural tube defect | 0 | 0 | 1 |
  Cardiac septal defect/murmur | 0 | 1 | 1 |
  Coarctation of aorta | 0 | 1 | 0 |
  Tetralogy of Fallot | 0 | 0 | 1 |
  Esophageal defects | 0 | 1 | 1 |
  Hypospadias | 1 | 0 | 0 |
  Hydroencephalopathy | 1 | 0 | 0 |
  Omphalocele | 0 | 1 | 0 |
  Extra digit | 0 | 0 | 1 |
  Skin tags on ear | 0 | 0 | 1 |

ADVERSE EVENTS:
Description: This was a prospective enrollment/follow-up study based on exposure/outcome data collected using structured enrollment and birth outcome report forms completed by healthcare providers of pregnant women. This observational study was designed to investigate birth defects, a specific group of serious adverse events (SAEs); no other SAEs were measured.
Groups:
- Lamotrigine Monotherapy Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine monotherapy with completed pregnancy outcome (does not include those lost to follow up where outcome information could not be obtained)
- Lamotrigine Polytherapy With Valproate Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine polytherapy with valproate exposures with completed pregnancy outcome (does not include those lost to follow up where outcome information could not be obtained)
- Lamotrigine Polytherapy Without Valproate Pregnancy Exposures: Prospectively enrolled pregnancies exposed to lamotrigine polytherapy without valproate exposures with completed pregnancy outcome (does not include those lost to follow up where outcome information could not be obtained)
Arm/Group | Lamotrigine Monotherapy Pregnancy Exposures | Lamotrigine Polytherapy With Valproate Pregnancy Exposures | Lamotrigine Polytherapy Without Valproate Pregnancy Exposures
Serious Adverse Events (participants affected / at risk) | 35/1776 | 16/171 | 12/497
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine Monotherapy Pregnancy Exposures (N=1776) | Lamotrigine Polytherapy With Valproate Pregnancy Exposures (N=171) | Lamotrigine Polytherapy Without Valproate Pregnancy Exposures (N=497)
Anencephaly (Congenital, familial and genetic disorders) | 3 | 0 | 0
Cardiac septal defect/murmur (Congenital, familial and genetic disorders) | 0 | 2 | 2
Club foot (Congenital, familial and genetic disorders) | 3 | 2 | 0
Coarctation of aorta (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital atresia of anus (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cortical dysplasis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Diaphragmatic hernia (Congenital, familial and genetic disorders) | 2 | 0 | 0
Epidermolysis bullosa (Congenital, familial and genetic disorders) | 1 | 0 | 0
Esophageal defects (Congenital, familial and genetic disorders) | 0 | 0 | 2
Gastroschisis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hip dislocation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocephalus/spina bifida (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hydroencephalopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydronephrosis (Congenital, familial and genetic disorders) | 2 | 0 | 0
Hypoplastic left heart/left ventricle hypoplasia (Congenital, familial and genetic disorders) | 2 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 2 | 0 | 1
Light spot across entire abdomen (Congenital, familial and genetic disorders) | 1 | 0 | 0
Meningomyelocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Microcephaly (Congenital, familial and genetic disorders) | 0 | 1 | 0
Minor heart defect, unspecified (Congenital, familial and genetic disorders) | 1 | 0 | 0
Neural tube defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Omphalocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Orofacial clefts (Congenital, familial and genetic disorders) | 2 | 3 | 0
Polydactyly (Congenital, familial and genetic disorders) | 2 | 1 | 1
Pulmonary stenosis (Congenital, familial and genetic disorders) | 1 | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 2 | 1 | 0
Renal defect (absent, polysystic, fluid on kidney) (Congenital, familial and genetic disorders) | 3 | 0 | 0
Skin tags on ear (Congenital, familial and genetic disorders) | 0 | 0 | 1
Tetralogy of Fallot (Congenital, familial and genetic disorders) | 0 | 0 | 1
Transposition of great vessels (Congenital, familial and genetic disorders) | 2 | 1 | 0
Ventricular hypoplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Ventricular septal defects (Congenital, familial and genetic disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.